CLINICAL TRIAL: NCT03507023
Title: Effect of the Combination of Polyphenols Derived From the Hibiscus Sabdariffa and Lippia Citriodora on Slightly Hypertensive or Type 1 Hypertensive Volunteers
Brief Title: Effect of Hibiscus and Lippia Extract on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital General Universitario Elche (Other); Monteloeder SL (Unknown)
Responsible Party: Principal Investigator, María Herranz-Lopez, Assistant Professor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UniversidadMHE_Met
Record Dates: First submitted 2018-03-16; First posted 2018-04-24 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): 2 capsules per day, each with 400 mg Cellulose microcrystalline, for 6 weeks.
  Interventions: Dietary Supplement: Placebo
- Dietetic Supplement Group (Experimental): 2 Capsules per day of Metabolaid® (each capsule contains 250 mg Metabolaid®, 150 mg cellulose microcrystalline), for 6 weeks.
  Interventions: Dietary Supplement: Metabolaid®

INTERVENTIONS:
Dietary Supplement: Metabolaid® — 500 mg per day, in fasting conditions.
  Arms: Dietetic Supplement Group
Dietary Supplement: Placebo — 500 mg per day, in fasting conditions.
  Arms: Placebo Control

SUMMARY:
Determine if a double-blind, randomized, placebo-controlled clinical intervention, based on a dietetic intervention and physical exercise, supplemented with a polyphenolic extract, decreases blood pressure in hypertensive volunteers.

DETAILED DESCRIPTION:
Slightly hypertensive individuals, before diagnosed with type 1 hypertension, are generally monitored by their physician and given dietetic and physical activity guidelines. The objective of this intervention is to prevent onset of a hypertensive pathologic condition. However, in many cases, this intervention is unsuccessful, and therefore the patient must follow-up with anti-hypertensive drugs.

Here, in the current study, the objective is to include a nutritional supplement in the intervention in order to increase the probability of success of the diet/exercise intervention. Previous studies with the supplement Metabolaid has shown the product to significantly decrease the blood pressure of slightly hypertensive individuals. It is estimated, based on the results of previous clinical studies, that the polyphenolic content of the nutritional supplement will reduce at least an additional 10% of the blood pressure of the patients undergoing a diet and exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Slight or type 1 hypertension with no pharmacological treatment, but with annual controls of the blood pressure

Exclusion Criteria:

* Minors (under 18 years of age)
* volunteers with high cardiovascular disease risk
* pharmacological treatment for blood pressure
* presence of any chronic disease/condition
* known allergies regarding the supplement and/or placebo

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Changes in Blood Pressure Measurement with respect to baseline | Continuous measurements for 24 hours, 1 day per week, total 6 weeks
  Using a continuous blood pressure monitor (BPro continuous blood pressure monitor, HealthStats)
Changes in Blood Pressure Measurement with respect to baseline | One measurement per day, 1 day per week, total 6 weeks
  Single Blood Pressure measurements, using the Omron M6 Comfort device

SECONDARY OUTCOMES:
Total Cholesterol | At the beginning and end of the intervention, total 6 weeks
  Blood Sampling in Fasting conditions, in mg/dl
HDL Cholesterol | At the beginning and end of the intervention, total 6 weeks
  Blood Sampling in Fasting conditions, in mg/dl
LDL Cholesterol | At the beginning and end of the intervention, total 6 weeks
  Blood Sampling in Fasting conditions, in mg/dl
Triglycerides | At the beginning and end of the intervention, total 6 weeks
  Blood Sampling in Fasting conditions, in mg/dl
Glucose | At the beginning and end of the intervention, total 6 weeks
  Blood Sampling in Fasting conditions, in mg/dl
Weight, using a weight scale | Once a week, for 6 weeks
  In kg
Height, using measuring tape | Once a week, for 6 weeks
  in cm
BMI, calculated based on Weight and Height | Once a week, for 6 weeks
  in kg/m^2
Waist Circumference, using a measuring tape | Once a week, for 6 weeks
  in cm
Hip Circumference, using a measuring tape | Once a week, for 6 weeks
  in cm
Waist/Hip Ratio | Once a week, for 6 weeks
  Calculated as indicator of obesity, based on Waist and Hip Circumference measurements
Physical Activity Assessment using the Stanford 7-days physical activity recall questionnaire | At baseline, 3 and 6 weeks
  Subjective assessment of physical activity using a validated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernandez de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No